CLINICAL TRIAL: NCT02449252
Title: Efficacy of Consolidative Involved-site Radiotherapy Following Effective Chemotherapy for Patients With Limited-stage Follicular Lymphoma: Wuhan University Cancer Center -NHL01 Trial
Brief Title: Efficacy of Consolidative Involved-site Radiotherapy for Patients With Limited-stage Follicular Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Di Deng, Director, Clinical Research, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUCC-NHL01 Trial
Record Dates: First submitted 2015-05-07; First posted 2015-05-20 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Follicular Lymphoma
Keywords: limited stage FL; Involved-site Radiotherapy; Chemotherapy
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ISRT group (Experimental): Six cycles chemotherapy (cyclophosphamide 750mg/square meter on day 1 + doxorubicin 50mg/square meter on day 1 + vincristine 1.4mg/square meter on day 1 (up to a maxomal dose of 2 mg) + prednisone 60mg/square meter on day 1 through 5, repeated at 21-day intervals).
  Consolidation involved-site radiotherapy (ISRT) following in patients with complete or partial response beginning 1 month after the last cycle of chemotherapy.
  Interventions: Radiation: Consolidation involved-site radiotherapy (ISRT); Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone
- IFRT group (Active Comparator): Six cycles chemotherapy (cyclophosphamide 750mg/square meter on day 1 + doxorubicin 50mg/square meter on day 1 + vincristine 1.4mg/square meter on day 1 (up to a maxomal dose of 2 mg) + prednisone 60mg/square meter on day 1 through 5, repeated at 21-day intervals).
  Consolidation involved-field radiotherapy (IFRT) following in patients with complete or partial response beginning 1 month after the last cycle of chemotherapy.
  Interventions: Radiation: Consolidation involved-field radiotherapy (IFRT); Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone

INTERVENTIONS:
Radiation: Consolidation involved-site radiotherapy (ISRT) — six cycles modern CHOP chemotherapy. Involved-site radiotherapy (ISRT) is based on defining the site of gross disease before chemotherapy, the GTV and using a CT-based volume with an expansion to form a CTV in the cranio-caudal direction.
  Involved-site radiotherapy (ISRT) is given in 24Gy~30Gy in 12~15 fractions of 2 Gy 5 days per week.
  Arms: ISRT group
Radiation: Consolidation involved-field radiotherapy (IFRT) — six cycles modern CHOP chemotherapy. Radiotherapy field of involved-field radiotherapy defined by CALGB is encompassed the prechemotherapy gross tumor.
  Involved-field RT (IFRT) is given in 24Gy~30Gy in 12~15 fractions of 2 Gy 5 days per week.
  Arms: IFRT group
Drug: cyclophosphamide — patients in both arms will be given cyclophosphamide chemotherapy.
Drug: doxorubicin — patients in both arms will be given cyclophosphamide chemotherapy.
Drug: vincristine — patients in both arms will be given cyclophosphamide chemotherapy.
Drug: prednisone — patients in both arms will be given cyclophosphamide chemotherapy.

SUMMARY:
Radiotherapy (RT) is an important option for patients with limited stage FL. The recommended approach for patients with limited stage FL by The National Comprehensive Cancer Network (NCCN) is 24Gy~30Gy consolidation RT following effective systemic therapy. There is no universal consensus for a ''standard'' RT field size in the treatment of limited stage FL. The involved-site radiotherapy (ISRT) has been treated effectively for these patients. However, the certain target volumes of ISRT need to be defined for patients with limited stage FL after effective chemotherapy.

DETAILED DESCRIPTION:
Follicular lymphoma (FL) is the second most common histology of non-Hodgkin's lymphoma and has significantly increased in incidence over the past three decades. FL, grade 1 or 2 has been recognized as having an indolent natural history with good long-term survival rates despite a high risk of recurrence. Approximately 25% of patients present with stage I or II disease (limited stage FL) at diagnosis, and their 10-year overall survival (OS) rate ranges from 52% to 79%. The treatment options include radiotherapy (RT) alone, immunotherapy ± chemotherapy, immunotherapy ± chemotherapy + RT, and even observation for selected patients. There were no differences in OS.

RT is an important option for patients with limited stage FL. Despite the evidence and these international guidelines' recommendation that primary RT has been considered the preferred treatment approach, RT alone remains worrisomely under used in the treatment of limited stage FL. The positive result that immediate RT was associated with improved disease-specific and overall survival (OS) in patients with stage I and II follicular lymphoma has been shown in SEER data. The OS and disease-free survival (DFS) at 15 years for limited stage FL treated with RT range from 40% to 66% and 40% to 49%, respectively. However, some controversies consider that the literature describing outcomes of early-stage follicular lymphoma treated with RT alone largely consists of retrospective accounts of selected patients from single institutions treated in an era before modern chemotherapy and staging procedures. For patients underwent rigorous staging with stage I FL, the results of The National LymphoCare Study show that progression-free survival (PFS) was significantly improved with either R-chemotherapy or systemic therapy + RT compared with patients receiving RT alone. The OS has no differences among the diverse treatment approaches in these patients. This result is also approved by several recent data both prospective study and retrospective analysis. So, it is questioned whether RT alone, which was the historical standard, is still the best choice for patients with limited stage FL. On combined-modality therapy (CMT) of limited stage FL, combined consolidation RT with brief modern CHOP or CHOP-like chemotherapy can improve the result of DFS though the OS failed to improvement. At the same time, a definitive radiation-dose study in indolent lymphoma from the British National Lymphoma Investigation shows that the 5-year freedom from local progression and OS have no difference either a radiation dose of 24 Gy or a dose of 40 to 45 Gy, respectively. Therefore, the recommended approach for patients with limited stage FL by the National Comprehensive Cancer Network (NCCN) is 24Gy~30Gy consolidation RT following effective systemic therapy. The main controversy focuses on the timing of RT, the combination between chemotherapy and RT and the ongoing reduction in radiation field size.

FL is generally considered an incurable disease and has a long-term outcomes of PFS and OS. Long-term complications related to RT among patients with early-stage FL should be focused as it emphasizes on Hodgkin's lymphoma (HL). In a British study of 2,456 patients with NHL, the relative risk (RR) of all malignancies were 1.3 per 10,000 person-years. The most common late non-neoplastic events were cardiac disease and infertility. In a study conducted by the European Organization for Research and Treatment of Cancer (EORTC), all late non-neoplastic events were observed in 46% of 757 patients at a median follow-up of 9.4 years after NHL treatment.

There is no universal consensus for a ''standard'' RT field size in the treatment of limited stage FL. The primary objective of reducing the RT field size is to lower rates of radiation-induced toxicity and radiation-induced second malignancy in long-term survivors without compromising disease control. Some previous studies show that involved-field RT (IFRT), involved regional RT (IRRT), and extended-field RT (EFRT) have similar survival outcomes. Even the radiotherapy field size is involved node RT (INRT). The retrospective results of Campbell et al show that the PFS was no significant difference for patients who received IRRT compared with patients who received INRT. Compared with the IRRT group, the smaller RT field size in the INRT group did not result in an increased risk of distant failure without infield or regional recurrence (38%vs 32%, respectively). However, the OS was inferior in the INRT group at 10 years (71% vs 59%). The underlying reason may relate to the absence of effective systemic therapy. Moreover, there is not the definition of CTV of RT in the research of Campbell et al. The planning target volume (PTV) of INRT in the research was also only added with physiologic movement and interfraction setup variation from gross target volume (GTV) which encompassed the sites of known disease.

It is necessary to design a prospective study with effective systemic therapy and the certain target volumes to evaluate the efficacy and adverse events of RT with smaller RT field size. Involved-site radiotherapy (ISRT), based on a modified involved field, aims to reduce the radiation volume treated and the probability of late effects. Its radiation targets include a gross tumor volume (GTV), a clinical target volume (CTV), and a planning target volume (PTV), which were defined in International Commission on Radiation Units and Measurements Report (ICRU) 50. This is based on defining the site of gross disease before chemotherapy, the GTV and using a CT-based volume with an expansion to form a CTV in the cranio-caudal direction.

Compared to the IFRT, the response rate and toxicities related to involved-site radiotherapy (ISRT) were to be evaluated for CR and PR patients with limited-stage FL after effective systemic treatment. The CTV of ISRT is defined as the region including the prechemotherapy volume of disease with 1.5 cm margin expanded cranio-caudally in the direction of potential lymphatic spread. The CTV should not extend into air in the transverse plane and should be limited in the involved lymph node region defined by the Cancer and Leukemia Group B (CALGB). The PTV is then extended from CTV by adding the necessary margin for setup error and organ motion.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female aged range from 18 years to 65 years.
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1.
* All patients had histologically confirmed Follicular lymphoma, grade 1 or 2.
* Limited-stage FL patients at newly diagnosed or recurrent without RT in initial management.
* Adequate organ function.
* Negative pregnancy test.
* Signed informed consent document on file.

Exclusion Criteria:

* Woman who were pregnant or lactating.
* With severe local infection or general infective disease.
* Primary lymphoma in special organ including cuticula, center never system, gastrointestinal tract, testicle, and lung.
* With other second primary malignancy except cutaneum carcinoma.
* Being or planning to participate in other study.
* Any patient who in the opinion of the investigator should not participate in the study.

Withdrawal Criteria:

* Patient are free to withdrawal completely from the study at any time upon request.
* Patient in the study may be stopped with the patient agreement at any time at the discretion of investigator.
* In-field progression on irradiation ongoing.
* Poor tolerability adverse events in the period of chemotherapy or irradiation after enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival - PFS | from the date of diagnosis to the date of treatment failure or death from any cause, whichever occurs first, Assessed up to 100 months.
  Treatment failure was defined as any recurrence of non-Hodgkin lymphoma.
Adverse events with grade 3 or 4 - AEs | The time from the day of treatment to the day of the first documented disease progression or death from any cause, Assessed up to 24 months.
  Toxicity was scored according to the toxicity scale of the National Cancer Institute Common Terminology Criteria for Adverse Events 3.0.

SECONDARY OUTCOMES:
Overall survival - OS | From the initial diagnosis of follicular lymphoma to death from any cause, Assessed up to 120 months.
Rate of in-field progression | From the start of RT to the first documented disease progression within the radiotherapy field, Assessed up to 120 months.
Rate of out-field progression | From the start of RT to the first documented disease progression outside the radiotherapy field, Assessed up to 120 months.
Rate of regional failure | From the start of RT to the first documented disease progression outside of ISRT field but within the involved region defined as CALGB, Assessed up to 120 months.

CONTACTS AND LOCATIONS:
Locations (1):
- DiDeng, Wuhan, Hubei, China